CLINICAL TRIAL: NCT05218369
Title: Effects of Immunomodulation With Interleukin-6 Antagonists on the Coagulation System in Critically-ill Covid-19 Patients
Brief Title: Interleukin-6 Antagonists in Critically-ill Covid-19 Patients
Acronym: HEMOCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 1405-3/2022/EÜIG
Record Dates: First submitted 2022-01-29; First posted 2022-02-01 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; Critical Illness
Keywords: severe COVID-19; interleukin-6 antagonist; ClotPro; viscoelastic hemostasis assay
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill COVID-19 patients: Patients in ICU due to critical COVID-19 infection, who receive early (within the first 24 hours, but no later than 48 hours after intubation) IL-6 antagonist therapy at the consultant's discretion.
  Interventions: Drug: IL6 Antagonist

INTERVENTIONS:
Drug: IL6 Antagonist — Patients will receive IL-6 antagonist therapy at the consultant's discretion.

SUMMARY:
The emerging SARS-COV2 virus has shed a new light on the cross-talks between the immune and the hemostatic system. In this study we aim to evaluate the dynamic change in coagulation caused by the modulation of the inflammatory response by interleukin-6 antagonist as assessed by viscoelastic methods in critically ill COVID-19 patients. Furthermore we try to draw attention to possible associations between the endothelial cell injury, inflammation and coagulation.

DETAILED DESCRIPTION:
The emerging SARS-COV2 virus has shed new light on the cross-talk between the immune and the hemostatic system. Pathophysiologically in COVID-19 infection the thrombo-inflammatory process is initiated by the host's exaggerated systemic inflammatory response, also called "dysregulated immune response" that activates both the inflammatory and the coagulation cascade directly by inflammatory mediators and indirectly by causing endothelial cell injury. These mechanisms altogether contribute to the imbalance of the hemostasis that is characterized by a procoagulant state.

In this multicenter prospective observational study, we aim to evaluate the dynamic change in coagulation as a result of immunomodulation by interleukin-6 antagonists in critically ill COVID-19 patients. We will assess the hemostatic system by a viscoelastic hemostasis assay (Clotpro, Haemonetics Corporation, Boston). Furthermore, we try to draw attention to possible associations between endothelial cell injury, inflammation, and coagulation. To compare these parameters we will draw blood for analysis before administration of IL-6 antagonist then 24h after, 48h after, and 7 days after.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old)
* Clinical diagnosis of SARS-CoV2 infection with rtPCR confirmation
* Disease severity with the indication of immunomodulation therapy with interleukin-6 antagonist: acute respiratory failure that requires invasive, noninvasive ventilation , or high flow nasal oxygen therapy with the following parameters: FiO2 > 0,4, flow > 30L/min and C Reactive Protein > 75 mg/L

Exclusion Criteria:

* The patient had previously been administered one of the following immunomodulating drug: anakinra, tocilizumab, sarilumab
* Presence of any condition or drug in the medical history that can lead to immunosuppression
* Suspicion of infection (active tuberculosis, bacterial, viral, fungal) or level of procalcitonine higher than 0,5 ng/ml at the enrollment of the patient
* Number of thrombocyte lower than 50 x 109 / L
* More than >120 hours passed between the admission to the ICU and the administration of interleukin-6 antagonist
* Administration of any of the following drugs the week before or during the study: fibrinolytic therapy, factor products (PCC, ATIII, FVIIa, FXIII), fibrinogen, desmopressin, tranexamic acid, blood products (FFP, thrombocyte concentrate)
* Pregnancy
* The patient or his legal guardian does not sign the consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to intensive care units (ICUs) requiring mechanical ventilation with proven COVID-19 infection and treated with interleukin-6 antagonist therapy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the lysis time | 48 hours
  Change of the fibrinolytic system before (T0) and after immunomodulation therapy, measured by the lysis time (LT).
Change in the lysis onset time | 48 hours
  Change of the fibrinolytic system before (T0) and after immunomodulation therapy, measured by the lysis onset time (LOT).

SECONDARY OUTCOMES:
Change in the lysis time | 24 hours and 7 days
  Change of the fibrinolytic system before (T0) and after immunomodulation therapy, measured by the lysis time (LT).
Change in the lysis onset time | 24 hours and 7 days
  Change of the fibrinolytic system before (T0) and after immunomodulation therapy, measured by the lysis onset time (LOT).
Change in Clotpro assay | 24 hours, 48 hours, and 7 days
  Change in blood coagulation parameters which evaluate hypercoagulable state before (T0) and after immunomodulation therapy (T1,2,3) measured by Clotpro device assays.
Correlation between procalcitonin and Clotpro | 24 hours, 48 hours, and 7 days
  Correlation between inflammatory and blood coagulation parameters. For the assessment of this endpoint, we will use the results of the inflammatory laboratory parameters as procalcitonin and the blood coagulation parameters measured by the Clotpro.
Correlation between C reactive protein and Clotpro | 24 hours, 48 hours, and 7 days
  Correlation between inflammatory and blood coagulation parameters. For the assessment of this endpoint, we will use the results of the inflammatory laboratory parameters as C reactive protein and the blood coagulation parameters measured by the Clotpro.
Correlation between ferritin and Clotpro | 24 hours, 48 hours, and 7 days
  Correlation between inflammatory and blood coagulation parameters. For the assessment of this endpoint, we will use the results of the inflammatory laboratory parameters as ferritin and the blood coagulation parameters measured by the Clotpro.
Correlation between lactate dehydrogenase and Clotpro | 24 hours, 48 hours, and 7 days
  Correlation between inflammatory and blood coagulation parameters. For the assessment of this endpoint, we will use the results of the inflammatory laboratory parameters as lactate dehydrogenase and the blood coagulation parameters measured by the Clotpro.
Correlation between syndecan-1 and Clotpro | 24 hours, 48 hours, and 7 days
  Correlation between biomarkers of endothelial injury and blood coagulation parameters. For the assessment of this endpoint, we will use the results of the biomarkers of the endothelial damage as syndecan-1 and the blood coagulation parameters measured by the Clotpro.
Correlation between thrombomodulin and Clotpro | 24 hours, 48 hours, and 7 days
  Correlation between biomarkers of endothelial injury and blood coagulation parameters. For the assessment of this endpoint, we will use the results of the biomarkers of the endothelial damage as thrombomodulin and the blood coagulation parameters measured by the Clotpro.

CONTACTS AND LOCATIONS:
Locations (3):
- Hungary (3):
  - Department of Anaesthesiology and Intensive Therapye, Medical School, University of Pécs, Pécs, Baranya
  - Central Department of Anesthesiology and Intensive Care, Szent György University Teaching Hospital of County Fejér, Székesfehérvár, Fejér
  - Department of Anaesthesiology and Intensive Therapy, Pest Megyei Flór Ferenc Hospital, Kistarcsa, Pest County

IPD SHARING:
Plan to Share IPD: No
Data will be presented at conferences and in the results part of the article.

REFERENCES:
- [Background] Gupta A, Madhavan MV, Sehgal K, Nair N, Mahajan S, Sehrawat TS, Bikdeli B, Ahluwalia N, Ausiello JC, Wan EY, Freedberg DE, Kirtane AJ, Parikh SA, Maurer MS, Nordvig AS, Accili D, Bathon JM, Mohan S, Bauer KA, Leon MB, Krumholz HM, Uriel N, Mehra MR, Elkind MSV, Stone GW, Schwartz A, Ho DD, Bilezikian JP, Landry DW. Extrapulmonary manifestations of COVID-19. Nat Med. 2020 Jul;26(7):1017-1032. doi: 10.1038/s41591-020-0968-3. Epub 2020 Jul 10. PMID 32651579
- [Background] Jackson SP, Darbousset R, Schoenwaelder SM. Thromboinflammation: challenges of therapeutically targeting coagulation and other host defense mechanisms. Blood. 2019 Feb 28;133(9):906-918. doi: 10.1182/blood-2018-11-882993. Epub 2019 Jan 14. PMID 30642917
- [Background] Levy JH, Iba T, Olson LB, Corey KM, Ghadimi K, Connors JM. COVID-19: Thrombosis, thromboinflammation, and anticoagulation considerations. Int J Lab Hematol. 2021 Jul;43 Suppl 1(Suppl 1):29-35. doi: 10.1111/ijlh.13500. PMID 34288441
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Levi M, Thachil J, Iba T, Levy JH. Coagulation abnormalities and thrombosis in patients with COVID-19. Lancet Haematol. 2020 Jun;7(6):e438-e440. doi: 10.1016/S2352-3026(20)30145-9. Epub 2020 May 11. No abstract available. PMID 32407672
- [Background] Bester J, Pretorius E. Effects of IL-1beta, IL-6 and IL-8 on erythrocytes, platelets and clot viscoelasticity. Sci Rep. 2016 Aug 26;6:32188. doi: 10.1038/srep32188. PMID 27561337
- [Background] Tleyjeh IM, Kashour Z, Damlaj M, Riaz M, Tlayjeh H, Altannir M, Altannir Y, Al-Tannir M, Tleyjeh R, Hassett L, Kashour T. Efficacy and safety of tocilizumab in COVID-19 patients: a living systematic review and meta-analysis. Clin Microbiol Infect. 2021 Feb;27(2):215-227. doi: 10.1016/j.cmi.2020.10.036. Epub 2020 Nov 5. PMID 33161150
- [Derived] Kovacs EH, Rottler M, Ruszkai Z, Gered C, Kiss T, Csata M, Reger B, Jakabfi-Csepregi R, Papp I, Turan C, Hegyi P, Fazakas J, Molnar Z, Tanczos K. Exploratory Analysis of Coagulation and Fibrinolysis Trajectories After IL-6 Antagonist Therapy in COVID-19: A Case Series. Biomedicines. 2026 Jan 22;14(1):254. doi: 10.3390/biomedicines14010254. PMID 41595788
- [Derived] Kovacs EH, Rottler M, Dembrovszky F, Ocskay K, Szabo L, Hegyi P, Molnar Z, Tanczos K. Investigating the association between IL-6 antagonist therapy and blood coagulation in critically ill patients with COVID-19: a protocol for a prospective, observational, multicentre study. BMJ Open. 2022 Nov 4;12(11):e063856. doi: 10.1136/bmjopen-2022-063856. PMID 36332964
- See also: Related Info — https://tm-centre.org/en/research/clinical-trials/